CLINICAL TRIAL: NCT05222399
Title: Pharmacokinetics of LY3871801 Following Oral Administration of a Crystalline Freebase Tablet and a Solid Dispersion Oral Suspension
Brief Title: A Study of LY3871801 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 18323; J3P-MC-FTAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3871801 (Period 1) (Experimental): LY3871801 solid dispersion suspension administered orally.
  Interventions: Drug: LY3871801
- LY3871801 (Period 2) (Experimental): LY3871801 crystalline freebase tablet administered orally.
  Interventions: Drug: LY3871801

INTERVENTIONS:
Drug: LY3871801 — Administered orally.

SUMMARY:
The main purpose of this study is to compare the amount of LY3871801 that gets into the blood stream and how long it takes the body to get rid of it, when given as crystalline freebase tablet (test) and as a solid dispersion oral suspension (reference) in healthy participants. The information about any adverse effects experienced will be collected and the tolerability of LY3871801 will also be evaluated. The study may last up to approximately 15 days excluding the 28 days of screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history and physical examination.
* Have body weight ≥ 45 kilograms (kg) and body mass index (BMI) within the range 18.5 to 40.0 kilograms per meter squared (kg/m²)
* Participants not of childbearing potential

Exclusion Criteria:

* Have known allergies to LY3871801, related compounds or any components of the formulation, or history of significant atopy.
* Have an abnormal blood pressure and/or pulse rate, deemed to be clinically significant by the investigator
* Have used or intend to use prescription or nonprescription medication (including dietary supplements, vitamins, herbal supplements, and/or alternative medicines) within 7 days prior to dosing
* History of drug or alcohol abuse in the past 2 years and/or regularly use known drugs of abuse
* Are unwilling to stop alcohol consumption 24 hours prior to admission and while resident at the clinical research unit (CRU).
* Smoke more than 10 cigarettes per day (or the equivalent, including electronic cigarettes) or are unable to abide by the CRU smoking restrictions.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3871801 | Predose through Day 4
  PK: Cmax of LY3871801
PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of LY3871801 | Predose through Day 4
  PK: AUC[0-∞] of LY3871801

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No